CLINICAL TRIAL: NCT05169801
Title: To Compare the Efficacy and Safety of BP102 in Combination With Paclitaxel/Carboplatin and Avastin® in Combination With Paclitaxel/Carboplatin in First-line Treatment of Advanced or Relapsed NSCLC - a Randomized, Double-blind, Positive Parallel Control, Multicentre Phase III Clinical Trial
Brief Title: To Compare the Efficacy and Safety of BP102 vs. Avastin® in Combination With Paclitaxel/Carboplatin in First-line Treatment of Advanced or Relapsed NSCLC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR-BP102-III-NSCLC
Record Dates: First submitted 2021-12-23; First posted 2021-12-27 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Non-small Cell Lung Cancer(NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Carboplatin; Bevacizumab

STUDY DESIGN:
Intervention Model Description: BP102 in combination with paclitaxel/carboplatin compared with Avastin® in combination with paclitaxel/carboplatin
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental)
  Interventions: Drug: BP102, paclitaxel, carboplatin
- Treatment group B (Active Comparator)
  Interventions: Drug: Avastin®, paclitaxel, carboplatin

INTERVENTIONS:
Drug: BP102, paclitaxel, carboplatin — BP102, paclitaxel, carboplatin
  Arms: Treatment group A
Drug: Avastin®, paclitaxel, carboplatin — Avastin®, paclitaxel, carboplatin
  Arms: Treatment group B

SUMMARY:
This is a randomized, double-blind, positive parallel control, multicentre Phase III clinical trial, a clinical trial of biosimilar drugs, so the type of comparison is equivalence test.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 18 to 75 (including 18 and 75), male or female;
2. Patients with locally advanced and unresectable NSCLC that has been histologically or cytologically proven, metastatic, or recurrent NSCLC.
3. No previous systematic antitumor therapy for current stage diseases. If previous adjuvant therapy has been received, it is necessary to ensure that the interval between the end of adjuvant therapy and the first administration of this study is more than 6 months, and that all adjuvant treating-related toxic reactions have recovered.
4. Patients must be able to document the EGFR mutation and ALK fusion gene status, and ALK must be negative. Patients who have not previously been tested for EGFR and ALK genes should be tested during screening;
5. There must be at least one measurable lesion as a target (according to RECIST V1.1);
6. ECOG: 0~1;
7. Life expectancy ≥24 weeks;
8. Major organs' function well.

Exclusion Criteria:

1. Patients with non-small cell lung cancer of other pathological tissue types;
2. Tumor histology or cytology confirmed positive ALK fusion gene;
3. Patients with imaging evidence of tumor invasion of large blood vessels;
4. Patients with uncontrolled pleural effusion and pericardial effusion that require repeated drainage;
5. Patients with abdominal effusion;
6. During the screening period, chest CT showed tumor cavity formation, or CT scan was highly suspected of idiopathic pulmonary fibrosis, mechanized pneumonia, drug-associated pneumonia, idiopathic pneumonia or active pneumonia;
7. Patients with hypertension whose blood pressure has not been satisfactorily controlled by antihypertensive drugs, and patients with previous hypertensive crisis or hypertensive encephalopathy;
8. Have heart disease or clinical symptoms that are not well controlled;
9. Patients with unhealed wounds, active gastric ulcers or fractures;
10. Patients diagnosed with esophagotracheal fistula;
11. People with known hereditary bleeding tendency or coagulation disorder;
12. Patients with known central nervous system metastases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2021-06-17 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 18 weeks
  optimal ORR at 18 weeks, independent radiographic assessment

SECONDARY OUTCOMES:
Progression-free survival | 41 months
  Progression-free survival is the time from randomization to the first documented objective disease progression (PD) using RECIST v1.1 or death due to any cause, whichever occurs first.
Overall survival (OS) | 41 months
  Overall survival is defined as the time from day 1 (part 1) or from randomization (part 2) to date of death.
Disease Control Rate (DCR) | 41 months
  Based on investigator reviewed radiographic tumour assessment and death.
Duration of Response (DoR) | 41 months
  Based on investigator reviewed radiographic tumour assessment and death.
Quality of Life assessment using EORTC QLQ-C30 | 41 months
  Evaluate subjects' quality of life
Incidence of treatment-emergent adverse events, serious adverse events | Enrollment to 28 days after permanent treatment termination
  Safety analyses will be performed using the safety population, defined as all patients receiving any study drug.
Positive rate of anti-bevacizumab antibody and its titer | 41 months
  Immunogenicity evaluation
Positive rate of neutralizing antibody | 41 months
  Immunogenicity evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Cancer Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided